CLINICAL TRIAL: NCT03975283
Title: Use of Long-acting Local Analgesia in Bariatrics: A Randomized Controlled Trial
Brief Title: Use of Exparel for Postoperative Analgesia Following Bariatric Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McMaster University (Other)
Collaborators: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SJHC80
Record Dates: First submitted 2019-05-31; First posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Injections; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Exparel (Liposomal Bupivicaine) (Experimental): 20 ml vial of liposomal bupivacaine containing 266 mg (maximum dose), will be diluted with 20 ml of 0.25% bupivacaine (containing 50 mg of bupivacaine) and 20 ml saline (60 ml total). That total volume will be divided into two 30 ml syringes, and each will be used (per side) for the TAP blocks.
  Interventions: Drug: Exparel 266 MG Per 20 ML Injection
- 0.25% Bupivicaine HCL (Active Comparator): Two 30 ml of 0.25% bupivacaine is drawn up and given on each side after identification of planes and levels via laparoscopy. Medication will be given just below the last rib and extend to below the lowest incision.
  Interventions: Drug: Bupivacaine Hcl 0.25% Inj

INTERVENTIONS:
Drug: Exparel 266 MG Per 20 ML Injection — 266mg of liposomal bupivacaine 266 mg, 20 mL volume, will be diluted with 20 ml of 0.25% bupivacaine (50 mg of bupivacaine) and 20 ml saline, thereby totalling 60mL volume. Total volume will be divided into two 30 ml syringes, and each will be used (per side) for the TAP blocks.
  Arms: Exparel (Liposomal Bupivicaine)
Drug: Bupivacaine Hcl 0.25% Inj — 0.25% bupivacaine, 60mL total, divided into two 30mL syringes and delivered via TAP block on either side.
  Arms: 0.25% Bupivicaine HCL

SUMMARY:
The aim of this study is to evaluate the efficacy of liposomal bupivicaine in post operative analgesia for patients undergoing bariatric surgery when compared to conventional local analgesia. Patients will be randomly selected to receive either liposomal bupivicaine or conventional bupivicaine via a transversus abdominal plane block during surgery. Patients will be followed post-operatively to assess use of narcotics, post-operative pain and nausea scores, and length of stay.

DETAILED DESCRIPTION:
Optimizing pain management following bariatric surgery is an important aspect of patient care and post-surgical recovery. Despite advances in post-operative pain management, this remains a challenge and opioids continue to dominate as the most widely used analgesia for post-surgical pain management. Opioid use especially in the opioid-naive patient carries significant short term and long term risks including over dependence and chronic opioid use.

Movements towards minimizing post-operative opioid use has shown regional anesthetic techniques to be highly effective in the management of pain in surgical patients. More specifically, liposomal bupivicaine (Exparel) is a novel non-opioid local analgesia that takes advantage of a multi-vesicular liposomal system to provide extended analgesia release over 72-96 hours.

The purpose of this study to evaluate the use of liposomal bupivicaine in the management of post-operative pain following bariatric surgery via a transversus abdominis plane (TAP) block. Patients will be randomized to receiving either liposomal bupivicaine or traditional 0.25% bupivicaine locally infiltrated at the time of bariatric surgery. Both liposomal bupivicaine and traditional bupivicaine will be administered via TAP block after identification of planes via laparoscopy by the bariatric surgeon.

Patients will be followed post-operatively to assess use of opioid analgesia between the two arms. In addition, they will be assessed with respect to pain and nausea using analog scores, as well as hospital length of stay.

ELIGIBILITY:
Inclusion Criteria:

* The patient previously met NIH criteria for bariatric surgery and has not received a previous bariatric surgical procedure
* The patient is aged 18-65 years and has completed the screening and preparation process prescribed by the Ontario Bariatric Network

Exclusion Criteria:

* Inability to give informed consent
* ASA > 4
* Planned procedure other than Roux-en-Y gastric bypass (RYGB) or contraindications to RYGB
* BMI > 55 kg/m2
* Revisional procedure
* Allergies or suspected allergies to local anesthetic medications (bupivicaine)
* Renal insufficiency (GFR < 30ml/min)
* History of chronic pain needing daily medications for the last >3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Efficacy of liposomal bupivicaine via TAP block in eliminating narcotic use post-operatively | 10 days
  Proportion of patients requiring narcotics post-procedure until discharge as recorded via their electronic medical record.

SECONDARY OUTCOMES:
Analog pain scores | 10 days (or until discharge)
  Pain will be assessed in the post-anaesthesia care unit (PACU) at 2 occasions - upon arrival and before transfer to ward. Subsequently, pain scores will then be reassessed at 8 am, 2 pm, and 8pm until discharge. Pain will be measured on an 11-point scale from 0 (no pain) to 10 (most pain imaginable) and the average of the PACU and ward scores will be used as the final outcomes.
Post-operative nausea | 10 days (or until discharge)
  Postoperative nausea scores will be assessed daily at 8 am, 2 pm, and 8pm until discharge using an 11-point scale from 0 (no nausea) to 10 (most nausea imaginable)
Post-operative Narcotic Use | 10 days (or until discharge)
  Postoperative narcotic use will be recorded in morphine equivalent units and recorded via their electronic medical record.
Hospital Length of Stay | Total length of stay will be calculated from registration until discharge to home; usually spans 2-5 days.
  Length of stay calculated in hours

CONTACTS AND LOCATIONS:
Overall Officials: Margherita Cadeddu, MD, FRCSC, Principal Investigator — McMaster University

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data

REFERENCES:
- [Background] Raebel MA, Newcomer SR, Bayliss EA, Boudreau D, DeBar L, Elliott TE, Ahmed AT, Pawloski PA, Fisher D, Toh S, Donahoo WT. Chronic opioid use emerging after bariatric surgery. Pharmacoepidemiol Drug Saf. 2014 Dec;23(12):1247-57. doi: 10.1002/pds.3625. Epub 2014 Apr 14. PMID 24733580
- [Background] Chahar P, Cummings KC 3rd. Liposomal bupivacaine: a review of a new bupivacaine formulation. J Pain Res. 2012;5:257-64. doi: 10.2147/JPR.S27894. Epub 2012 Aug 14. PMID 23049275
- [Background] Dasta J, Ramamoorthy S, Patou G, Sinatra R. Bupivacaine liposome injectable suspension compared with bupivacaine HCl for the reduction of opioid burden in the postsurgical setting. Curr Med Res Opin. 2012 Oct;28(10):1609-15. doi: 10.1185/03007995.2012.721760. Epub 2012 Sep 3. PMID 22900785
- [Background] Cohen SM. Extended pain relief trial utilizing infiltration of Exparel((R)), a long-acting multivesicular liposome formulation of bupivacaine: a Phase IV health economic trial in adult patients undergoing open colectomy. J Pain Res. 2012;5:567-72. doi: 10.2147/JPR.S38621. Epub 2012 Nov 20. PMID 23204866
- [Background] Bhakta A, Glotzer O, Ata A, Tafen M, Stain SC, Singh PT. Analgesic efficacy of laparoscopic-guided transverse abdominis plane block using liposomal bupivacaine in bariatric surgery. Am J Surg. 2018 Apr;215(4):643-646. doi: 10.1016/j.amjsurg.2017.09.006. Epub 2017 Sep 20. PMID 29061282
- [Background] Boerboom SL, de Haes A, Vd Wetering L, Aarts EO, Janssen IMC, Geurts JW, Kamphuis ET. Preperitoneal Bupivacaine Infiltration Reduces Postoperative Opioid Consumption, Acute Pain, and Chronic Postsurgical Pain After Bariatric Surgery: a Randomized Controlled Trial. Obes Surg. 2018 Oct;28(10):3102-3110. doi: 10.1007/s11695-018-3341-6. PMID 29926357
- [Background] Ilfeld BM, Viscusi ER, Hadzic A, Minkowitz HS, Morren MD, Lookabaugh J, Joshi GP. Safety and Side Effect Profile of Liposome Bupivacaine (Exparel) in Peripheral Nerve Blocks. Reg Anesth Pain Med. 2015 Sep-Oct;40(5):572-82. doi: 10.1097/AAP.0000000000000283. PMID 26204387
- [Background] Surdam JW, Licini DJ, Baynes NT, Arce BR. The use of exparel (liposomal bupivacaine) to manage postoperative pain in unilateral total knee arthroplasty patients. J Arthroplasty. 2015 Feb;30(2):325-9. doi: 10.1016/j.arth.2014.09.004. Epub 2014 Sep 16. PMID 25282071
- [Background] Bramlett K, Onel E, Viscusi ER, Jones K. A randomized, double-blind, dose-ranging study comparing wound infiltration of DepoFoam bupivacaine, an extended-release liposomal bupivacaine, to bupivacaine HCl for postsurgical analgesia in total knee arthroplasty. Knee. 2012 Oct;19(5):530-6. doi: 10.1016/j.knee.2011.12.004. Epub 2012 Jan 28. PMID 22285545
- [Background] Ilfeld BM, Malhotra N, Furnish TJ, Donohue MC, Madison SJ. Liposomal bupivacaine as a single-injection peripheral nerve block: a dose-response study. Anesth Analg. 2013 Nov;117(5):1248-56. doi: 10.1213/ANE.0b013e31829cc6ae. PMID 24108252